CLINICAL TRIAL: NCT04655508
Title: Efficacy of Fluticasone Propionate Associated With Salmeterol Using Inhalation Chamber Versus Placebo to Improve the Respiratory Function in Children Over Six Years of Age Who Underwent Allogeneic Hematopoietic Stem Cell Transplantation With a Decline of FEV1 ≥10% From Pre Transplantation
Acronym: RESPPEDOBS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient enrollment.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP180600
Record Dates: First submitted 2020-11-10; First posted 2020-12-07 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-02

CONDITIONS: Stem Cell Transplant Complications; Respiratory Disease; Bronchiolitis Obliterans
MeSH Terms: conditions — Respiration Disorders; Bronchiolitis Obliterans | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Seretide (Experimental): For children between 6 to 11 years (< 12 years): 50 μg inhaled fluticasone propionate and 25 μg salmeterol (SERETIDE® 50/25) :two puffs twice a day from randomisation during 6 months using inhalation chamber
  - For children between 12 to 17 years (> or = 12 years) : 125 μg inhaled fluticasone propionate and 25 μg salmeterol (SERETIDE® 125/25): two puffs twice a day from randomisation during 6 months using inhalation chamber
  Interventions: Drug: Seretide
- placebo (Placebo Comparator): For children between 6 to 11 years (< 12 years): placebo of SERETIDE® 50/25 :two puffs twice a day from randomisation during 6 months using inhalation chamber For children between 12 to 17 years (> or = 12 years) : placebo of SERETIDE® 125/25: two puffs twice a day from randomisation during 6 months using inhalation chamber
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seretide — For children between 6 to 11 years (< 12 years): 50 μg inhaled fluticasone propionate and 25 μg salmeterol (SERETIDE® 50/25) :two puffs twice a day from randomisation during 6 months using inhalation chamber
  - For children between 12 to 17 years (> or = 12 years) : 125 μg inhaled fluticasone propionate and 25 μg salmeterol (SERETIDE® 125/25): two puffs twice a day from randomisation during 6 months using inhalation chamber
  Arms: Seretide
Drug: Placebo — For children between 6 to 11 years (< 12 years): placebo of SERETIDE® 50/25 :two puffs twice a day from randomisation during 6 months using inhalation chamber For children between 12 to 17 years (> or = 12 years) : placebo of SERETIDE® 125/25: two puffs twice a day from randomisation during 6 months using inhalation chamber
  Arms: placebo

SUMMARY:
Bronchiolitis Obliterative Syndrome (BOS) is the primary noninfectious pulmonary complication after hematopoietic stem cell transplantation (HSCT) and usually carries a poor prognosis. It occurs in about 10% of children underwent HSCT. The National Institutes of Health (NIH) published guidelines and criteria for the diagnosis of BOS. BOS defined by spirometric criteria according to modified NIH consensus guidelines: FEV1 < 75% predicted and a greater than 10% decline from pretransplant baseline, and FEV1/FVC <0.7 (FCV: Forced Vital Capacity). Nevertheless Cheng and al. indicate that the magnitude of FEV1 decline before diagnosis exceeded the diagnostic requirement of a greater than 10% decline compared with baseline FEV. Moreover, the decline in FEV1 prior to BOS diagnosis appeared to occur within 6 months for those patients. Recent studies suggest that any intervention should be targeted during the FEV1 decline, and before the diagnosis of BOS. For this, inhalated treatment are used: Bergeron et al. reported improvements in symptoms as well in FEV1 one month followed treatment including formoterol and budesonide in a prospective trial including adults (12% increase of FEV1 for 62% adults). Williams and al. in another prospective adult's cohort, showed that the association between fluticasone, montelukast and azythromycin was associated with stable lung function, reduced systemic corticosteroids, and improved quality of life at 3 months for adults with BOS.

In our national French prospective cohort which include 300 children with HSCT from 2014 to 2017 (RESPPEDHEM Programme Hospitalier de Recherche Clinique 2012), 35% of children presented a decline of FEV1≥ 10% without BOS criteria (FEV1 < 75% and FEV1/FVC <0.7). Among them, some received combination of corticoids and long acting beta agonists for 6 months. Children with this type of inhalated treatment improved their FEV1 to 88.1% predicted while children without any treatment have a FEV1 at 80.7% predicted. Our hypothesis is that association of Fluticasone Propionate and Salmeterol can be used as a treatment of the decline of FEV1 for children and so prevent BOS.

DETAILED DESCRIPTION:
It's a prospective randomized double blind, multicentre, parallel-group in a 1:1 ratio, controlled and superiority trial.

The primary objective is to assess the effect of a Fluticasone Propionate associated with Salmeterol using inhalation chamber compared to placebo on respiratory function at 6 months in children over six years of age who underwent allogeneic hematopoietic stem cell transplantation with a decline of FEV1 ≥ 10% from pre transplantation.

The primary criterion will be the difference in the FEV1% predicted value from inclusion to 6 months following the initiation of treatment.

To assess the effect of a Fluticasone Propionate associated with Salmeterol using inhalation chamber compared to placebo in children over six years old underwent allogeneic hematopoietic stem cell transplantation with a decline of FEV1 ≥ 10% from pre transplantation baseline to 6 months following the initiation of treatment, and 6 months after the end of treatment, on pulmonary function, respiratory symptoms, Bronchiolitis Obliterative Syndrome (BOS) rate, oral steroid exposure and occurrence of infections;

To assess potential confounding factors associated to the 6-months inhaled treatment efficacy from baseline to 12 months, especially:

- GVHD (Graft Versus Host Disease) occurrence, severity and treatment (steroid dose exposure, calcineurins inhibitors dose, second line of GVHD treatment); To assess the safety and tolerability of the treatment at baseline, M1, M3 and M6 following the initiation of treatment

All endpoints were collected at baseline, randomization, 1, 3, 6 months during the treatment period, and then 3, 6 months after the end of the treatment.

1. Endpoints relative to respiratory symptoms :

   * dyspnea will be evaluate at the NYHA (New York Heart Association) scoring;
   * step test (patient climb up and down step during three minutes at the frequency of 30/mn) : Respiratory rate, dyspnea Heart rate, SaO2 (oxygen saturation) during the exercise.
2. Endpoints relative to pulmonary function :

   * FEV1 (Forced expiratory volume) VC (Vital Capacity) , TLC (Total Lung capacity) , RV (Residual volume), FRC (Functional Residual Capacity), sRaw (specific airway resistance) DLCO (diffusing capacity of the lungs) using a similar method of measurement for static lung volumes (plethysmography)
   * Number of patients presented with BOS defined as the absence of infection, and FEV1 < 75% predicted, and the FEV1/ FVC < 0.7, and the RV >120% or air trapping or bronchiectasis or small airways thickening on computed tomography
3. Endpoints relative to GVHD :

   * Acute and Chronic GVHD manifestations defined on NIH consensus with scoring;
   * First line of treatment: cumulative dose of corticosteroid systemic exposure and cumulative dose of calcineurins inhibitors.
   * Second line of GVHD treatment exposure will be assessed using the other type of treatment.
4. Endpoints relative to respiratory infections :

   - Number of adverse events.
5. Endpoints relative to safety and tolerance:

   * Adverse events during the study period such as treatment tolerance, thrush, death.

The investigators will study patients over six years of age who underwent allogeneic hematopoietic stem cell transplantation with a decline of FEV1 ≥10% from pre transplantation.

The choice of this range of age is motivated by the fact that PFTs (Pulmonary Function Test) requires a degree of cooperation that is age dependent, only children who are 6 years of age or older are able to realize reproducible PFTs.

For children between 6 to 11 years (< 12 years): 50 μg inhaled fluticasone propionate and 25 μg salmeterol (SERETIDE® 50/25) :two puffs twice a day from randomisation during 6 months using inhalation chamber

- For children between 12 to 17 years (> or = 12 years) : 125 μg inhaled fluticasone propionate and 25 μg salmeterol (SERETIDE® 125/25): two puffs twice a day from randomisation during 6 months using inhalation chamber For children between 6 to 11 years (< 12 years): placebo of SERETIDE® 50/25 :two puffs twice a day from randomisation during 6 months using inhalation chamber For children between 12 to 17 years (> or = 12 years) : placebo of SERETIDE® 125/25: two puffs twice a day from randomisation during 6 months using inhalation chamber

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescent aged 6 to 17 years
* Getting an Allo Hematopoietic cell stem transplantation
* Provide written informed consent from legal guardian
* Covered by medical insurance (social security ou CMU).

Randomisation criteria:

- Decline of FEV1 ≥ 10% from pre transplantation between M3 and M12 after the transplantation, confirmed over two functional test performed one week apart, without Bronchiolitis Obliterative Syndrome international criteria, neither initiation of inhaled treatment from transplantation to randomization visit.

Exclusion Criteria:

* Patients with no affiliation to a social security scheme (beneficiary or legal)
* Pregnancy
* Asthma defined by reversibility with salbutamol (FEV1 > 12% or FEV1> 200ml) under inhaled corticosteroids or long acting beta agonists during the last three months
* Patients with hypersensitivity to the active substances: salmeterol, fluticasone propionate, or to the excipients: norflurane.

Non-Randomisation criteria :

* Viral respiratory infection (fever ≥ 38°C, tachypnea according to age, positive viral PCR (Polymerase Chain Reaction) pharyngeal aspiration) during the last month;
* Lower respiratory tract infection (fever ≥ 38°C, tachypnea, radiologically or echography confirmed pneumonia, sputum) during the last month;
* Invasive fungal disease (as defined by European Organisation for Research and Treatment of Cancer/Mycoses Study Group consensus group) during the last month.
* Potent cytochrome P450 3A4 inhibitors, such as ritonavir, ketoconazole, itraconazole, troleandomycin, clarithromycin, nelfinavir and nefazodone.
* Corticosteroids or bronchodilatators inhaled treatment after transplantation
* Bronchiolitis Obliterative Syndrome

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
FEV: Forced Expiratory Volume in 1 second | The primary criterion will be measured at months 0, 1, 3, 6, 9 and 12.
  The primary criterion will be the change in the FEV1% predicted value from inclusion to 6 months following the initiation of treatment

SECONDARY OUTCOMES:
Graft Versus Host Disease | The criterion will be measured at months 0, 1, 3, 6, 9 and 12.
  GVHD occurrence (Acute and Chronic GVHD manifestations defined on NIH consensus with scoring), First line of treatment: cumulative dose of corticosteroid systemic exposure and cumulative dose of calcineurins inhibitors and Second line of GVHD treatment exposure will be assessed using the other type of treatment
Dyspnea | The criterion will be measured at months 0, 1, 3, 6, 9 and 12.
  dyspnea will be evaluate at the NYHA scoring from I to IV (I: none, IV: symptomatic at rest)
Step Test | The criterion will be measured at months 0, 1, 3, 6, 9 and 12.
  step test: Respiratory rate, dyspnea Heart rate, SaO2 during the exercise.
Bronchiolitis Obliterative Syndrome | The criterion will be measured at months 0, 1, 3, 6, 9 and 12.
  The investigators will measure the number of patients presented with Bronchiolitis Obliterative Syndrome
Adverse events | The criterion will be measured at months 0, 1, 3, 6, 9 and 12.
  The investigators will measure the Occurrence of infections
Pulmonary function | FEV1 will be measured at months 0, 1, 3, 6, 9 and 12
  A plethysmography will be performed to measured pulmonary parameters: FEV1 (Forced Expiratory Volume)
Pulmonary function | VC will be measured at months 0, 1, 3, 6, 9 and 12
  A plethysmography will be performed to measured pulmonary parameters: VC (Vital Capacity)
Pulmonary function | TLC will be measured at months 0, 1, 3, 6, 9 and 12
  A plethysmography will be performed to measured pulmonary parameters: TLC (Total Lung Capacity)
Pulmonary function | RV will be measured at months 0, 1, 3, 6, 9 and 12
  A plethysmography will be performed to measured pulmonary parameters: RV (Residual Volume)
Pulmonary function | FRC will be measured at months 0, 1, 3, 6, 9 and 12
  A plethysmography will be performed to measured pulmonary parameters: FRC (Functional Residual Capacity)
Pulmonary function | sRaw will be measured at months 0, 1, 3, 6, 9 and 12
  A plethysmography will be performed to measured pulmonary parameters: sRaw (Specific airway resistance)
Pulmonary function | DLCO will be measured at months 0, 1, 3, 6, 9 and 12
  A plethysmography will be performed to measured pulmonary parameters: DLCO (Diffusing Capacity of the Lungs)

CONTACTS AND LOCATIONS:
Locations (1):
- Houdouin véronique, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided